CLINICAL TRIAL: NCT01571011
Title: Chicago Urban Resiliency Building (CURB): Phase 3 Clinical Trial in Primary Care to Engage Adolescents With a Web-based Depression Prevention Intervention
Brief Title: Chicago Urban Resiliency Building (CURB)
Acronym: CURB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Van Voorhees, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Benjamin Van Voorhees, MD, MPH, Associate Professor of Pediatrics; Chief, Section of General Pediatrics and Adolescent Medicine; Director, TIKES Center Department of Pediatrics, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RWJF 68177
Record Dates: First submitted 2012-03-20; First posted 2012-04-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Major Depression
Keywords: Adolescent; Randomized Trial; Internet; Depressive Disorder; Primary Care; Prevention
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CURB Intervention (Experimental): The intervention is made up of 14 internet modules based on behavioral activation, cognitive behavioral therapy, and interpersonal psychotherapy as well as motivational interviews in the primary care setting (to enhance behavior change). It is suggested that an adolescent navigates through 2 modules a week. The motivational interviews with the physicians occur directly before and after the adolescent is exposed to the website (at baseline and 3 months) in the providers office. The parents of the enrolled adolescents are also invited to navigate through their own, 3 module, parent internet program.
  Interventions: Behavioral: CURB
- CURB Intervention (Wait List) (Experimental): Same as the CURB Intervention arm, however, individuals assigned to this arm wait 3 months before receiving the intervention.
  Interventions: Behavioral: CURB

INTERVENTIONS:
Behavioral: CURB — The intervention is made up of 14 internet modules based on behavioral activation, cognitive behavioral therapy, and interpersonal psychotherapy as well as motivational interviews in the primary care setting (to enhance behavior change). It is suggested that an adolescent navigates through 2 modules a week. The motivational interviews with the physicians occur directly before and after the adolescent is exposed to the website (at baseline and 3 months) in the providers office. The parents of the enrolled adolescents are also invited to navigate through their own, 3 module, parent internet program.

SUMMARY:
The purpose of the study is to determine whether a culturally tailored, low-cost, primary care/internet based depression prevention intervention (CURB) is superior to wait-list control for African American and Hispanic youth in terms of depression-related outcomes. It is hypothesized that compared to teens in the wait-list control condition, teens in the CURB program will exhibit lower levels of depressed mood and/or more rapid changes in mood during the follow-up time.

DETAILED DESCRIPTION:
Additional aims and hypotheses are provided here:

Aim 2: To determine whether or not participants in the CURB primary care/Internet based depression prevention intervention will have a significantly lower cumulative incidence of any depressive episode at 3 months compared to adolescents in the usual care wait-list group.

Hypothesis 2: Compared to youth in the wait-list control condition, youth in the CURB program will have a lower incidence of depressive episodes at 6 month follow-up.

Aim 3: To determine whether CURB is sustainable in primary care from the perspective of health care professionals and primary care physicians in urban primary care settings.

Hypothesis 3: We hypothesize that providers will rate the intervention (by component) feasibility, acceptability, willingness to perform intervention and sustainability > 7 on a 1-10 scale (1, not feasible, 10 very feasible).

ELIGIBILITY:
Inclusion Criteria:

Adolescents:

* Male and female African American and Latino/a youth ages 13 -17 years old.
* Adolescents with depressed mood (> 2 weeks duration) will be eligible unless they have already exceeded the diagnostic threshold for major depressive disorder or have a comorbid condition as defined in the exclusion criteria.

Parents:

* Parent of eligible adolescents

Primary Care Physicians (PCPs):

* Physician at one of the four Mile Square Health Centers.

Health Care Professionals:

* Employee at one of the four Mile Square Health Centers.

Exclusion Criteria:

* Adolescents undergoing active treatment for depression [Active treatment for depression is defined as receiving anti-depressant medication or counseling within one year of remission of symptoms from the most recent episode]
* Adolescents meeting probable diagnostic criteria for the following: Major depression, Substance and alcohol abuse, Panic attacks, Generalized anxiety disorder, Eating disorders, History of treatment for bi-polar disorder or schizophrenia or who are at elevated risk for suicide (often have suicidal thoughts or recent intent)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The Center for Epidemiological Studies of Depression (CES-D) Scale | 0, 3, 6 months
  Change in CESD from baseline Change in CESD scale between and within groups across the 6 months and for each assessment point

SECONDARY OUTCOMES:
Cost effective outcome measures | 6 months
Vulnerability | 6 months
Protective factors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Voorhees, MD, MPH, Principal Investigator — University of Illinois at Chicago; Monika Marko, MSS, Study Director — UIS
Locations (1):
- Mile Square Health Centers, Chicago, Illinois, United States

REFERENCES:
- See also: Sponsor — http://www.solvingdisparities.org/